CLINICAL TRIAL: NCT05652192
Title: Stereotactic Body Radiotherapy (SBRT) Combined With Chemotherapy and Tislelizumab in Metastatic Nasopharyngeal Carcinoma: A Single-arm, Phase Ⅱ Study
Brief Title: SBRT Combined With Chemotherapy and Tislelizumab in Metastatic NPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2022-514
Record Dates: First submitted 2022-11-08; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Advanced Nasopharyngeal Carcinoma

STUDY DESIGN:
Intervention Model Description: SBRT for metastatic diseases combined with systemic therapy with GP chemotherapy plus PD-1 antibody
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): SBRT: Metastases were treated with SBRT, GTV 45Gy/3F/3d, each course of radiotherapy only treated metastases within 1 organ.
  Chemotherapy(GP or TP) was combined with tislelizumab for 4-6 cycles and tislelizumab was maintained until 2 years or disease progression or intolerable toxicity or death.
  Maintain: (1) For newly diagnosed metastatic patients, nasopharyngeal and metastatic lymph node irradiation was started 4 weeks after systemic therapy, using IMRT technique, only radiating the GTV of the nasopharyngeal and cervical region, DT 66 Gy/30 F/6 weeks was recommended. Tislelizumab was continued during radiotherapy and tislelizumab was used during maintenance.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — SBRT was added to systematic treatment (chemo+ PD-1 antibody)

SUMMARY:
Radiotherapy and immunotherapy have achieved good survival benefit in advanced nasopharyngeal carcinoma. A number of clinical studies of immunotherapy combined with radiotherapy for nasopharyngeal carcinoma are also ongoing. This study preliminarily explored the efficacy and safety of SBRT combined with tislelizumab and chemotherapy in metastatic nasopharyngeal carcinoma. Hypofractionated radiotherapy combine with systemic chemotherapy and immunotherapy in advanced nasopharyngeal carcinoma. Not only it can achieve rapid response of distant metastases, but also to achieve long-term survival benefit for patients, which provides the reference for subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed a written informed consent form (ICF) voluntarily.
2. Male or female, aged from 18 to 75 years.
3. Pathologically confirmed newly diagnosed or treated metastatic patients are not suitable for radiotherapy.
4. Have not received treatment for metastatic nasopharyngeal carcinoma.
5. At least one metastatic lesion can be treated with SBRT.
6. ECOG score 0-1.
7. Expected survival expectancy of no less than 6 months.
8. Adequate bone marrow/liver and kidney function/heart and lung and other physiological function reserves, expected to successfully complete chemoradiotherapy and immunotherapy.
9. Women of childbearing potential must confirm a negative serum pregnancy test and agree to use effective contraception during study drug use and for 150 days after the last dose.
10. Male patients with sexual partners of childbearing potential must agree to use effective contraception during study drug use and for 150 days after the last dose. Subject is willing and able to comply with visits, treatment regimen, laboratory tests, and other requirements of the study as specified in the schedule.
11. Subjects are willing and able to comply with visits, treatment regimens, laboratory tests, and other requirements of the study as spe

Exclusion Criteria:

* 1. subjects with pathologically diagnosed adenocarcinoma or sarcoma of the nasopharynx.

  2. subject has other malignancy within 3 years prior to first dose except nasopharyngeal carcinoma. Subjects with other malignancies that have been cured by local therapy, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, cervical or breast carcinoma in situ, are excluded.

  3. Participated in treatment with an investigational drug or used an investigational device within 4 weeks prior to the first dose.

  4. Active autoimmune disease requiring systemic treatment within 2 years prior to the first dose, or autoimmune disease that may recur or plan treatment as judged by the investigator.

  5. active or previous definite inflammatory bowel disease (e.g., Crohn 's disease or ulcerative colitis) disease.

  6. History of immunodeficiency; positive HIV antibody test; current chronic use of systemic corticosteroids or other immunosuppressive agents; local, ocular, intra-articular, intranasal, and inhaled corticosteroids are allowed.

  7. Subjects with known active pulmonary tuberculosis (TB) and suspected active TB require clinical examination to rule out; known active syphilis infection.

  8. known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation; 9. history of pneumonitis/interstitial lung disease requiring systemic corticosteroids or current pneumonitis.

  10. serious infections within 4 weeks prior to the first dose, including but not limited to comorbidities requiring hospitalization, sepsis, or serious pneumonia; active infections (excluding antiviral therapy for hepatitis B or C) that have received systemic anti-infective therapy within 2 weeks prior to the first dose.

  11. Subjects with untreated active hepatitis B (HBsAg positive and HBV-DNA more than 1000 copies/ml [200 IU/ml] or above the lower limit of detection) and anti-hepatitis B virus treatment during study treatment are required for subjects with hepatitis B; subjects with active hepatitis C (HCV antibody positive and HCV-RNA level above the lower limit of detection).

  12. any of the following cardiovascular and cerebrovascular diseases: a) myocardial infarction, unstable angina pectoris, cerebrovascular accident, transient ischemic attack, acute or persistent myocardial ischemia, symptomatic heart failure (Grade 2 and above according to the New York Heart Association functional classification), or any arterial thromboembolic event within 6 months before the first dose; b) history of venous thromboembolic events (NCI CTCAE 5.0 version 3 and above), pulmonary embolism, or other serious thromboembolism within 3 months before the first dose; c) presence of serious arrhythmia requiring long-term drug intervention; patients with asymptomatic atrial fibrillation with stable ventricular rate are allowed; d) presence of aortic aneurysm, aortic dissecting aneurysm, internal carotid artery stenosis and other major vascular diseases that may be life-threatening or require surgery within 6 months; e) previous history of myocarditis or cardiomyopathy.

  13. Known hypersensitivity to any component of any study drug; known history of serious hypersensitivity to other monoclonal antibodies.

  14. known history of mental illness, drug abuse, alcoholism, or drug abuse; 15. pregnant or lactating women. 16. Any previous or current illness, treatment, or laboratory abnormality that may confound the results of the study, affect the subject 's full participation in the study, or that participation may not be in the subject' s best interest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 years

SECONDARY OUTCOMES:
ORR | 2 years
  target lesion objective response rate after SBRT and 4-6 cycle chemo +immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: feng Jiang, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No